CLINICAL TRIAL: NCT05000502
Title: Exercise, Gut Microbiome, and Breast Cancer: Increasing Reach to Underserved Populations
Acronym: EMBRACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Laura Q. Rogers, MD, MPH, Professor, Med - Preventive Medicine, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 300007016; BCRFA (Other: Breast Cancer Research Foundation of Alabama)
Record Dates: First submitted 2021-08-03; First posted 2021-08-11 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Female Breast Cancer
Keywords: Exercise; Gut Microbiome; Breast Cancer; Cancer; Aerobic Exercise; Microbiome; Female Breast Cancer; Flexibility Exercise
MeSH Terms: conditions — Motor Activity; Breast Neoplasms; Neoplasms

STUDY DESIGN:
Intervention Model Description: 40 breast cancer survivors will be randomized (like flipping a coin) to one of two study conditions: 1) home-based aerobic exercise training (with aerobic exercise progression targeting improved cardiorespiratory fitness) or 2) standard attention control (stretching exercises). All participants will be asked to maintain their usual diet and avoid change in body weight during the study.
Who Masked: Outcomes Assessor
Masking Description: Staff doing assessments will be masked to study group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-based aerobic exercise training (Experimental): home-based aerobic exercise condition will receive a fitness bracelet (with heart rate measurement capability) and weekly exercise counseling from an exercise trainer (i.e., exercise physiologist) by videoconference. The weekly counseling will be guided by the fitness bracelet data (both participant and exercise trainer will share the same log in information). The aerobic exercise progression will gradually increase duration and intensity of aerobic exercise with the goal of improving cardiorespiratory fitness.
  Interventions: Behavioral: Home-based exercise intervention
- Home-based standard attention flexibility/toning control (Active Comparator): Home-based standard attention flexibility/toning control will receive light resistance bands, stretching/toning log book, and weekly videoconference counseling from an exercise trainer.
  Interventions: Behavioral: Home-based exercise intervention

INTERVENTIONS:
Behavioral: Home-based exercise intervention — A 10-week home-based exercise intervention including weekly video conferences with exercise specialists.

SUMMARY:
Understanding the impact exercise has on a cancer survivor's gut microbiome can improve the health and well-being of cancer survivors by enhancing treatments targeting the gut microbiome. Although scientific studies support a link between exercise and the gut microbiome, rigorous randomized trials needed to confirm this causal link are limited and usually involve supervised exercise. Hence, this proposal tests feasibility of a home-based, remote-only research protocol that is more accessible to cancer survivors unable to attend supervised exercise including but not limited to rural populations. This study will also determine if exercise effects on the gut microbiome differ by factors such as race.

DETAILED DESCRIPTION:
Forty physically inactive breast cancer survivors will be randomized into 10-week conditions of home-based aerobic exercise training or standard attention control. All participants will be asked to maintain their pre-study diet and attempt to maintain their body weight while participating in the study. Assessments will occur at baseline, week 5 (mid-intervention), and week 10 (post-intervention) by videoconference platform. Study feasibility and changes in the gut microbiome will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Non-Hispanic white or black women
* Age 18-70 years
* History of breast cancer stage 0, I, II, or III
* ≥1 year post-primary cancer treatment completion
* English speaking
* Ambulates without assistance
* No antibiotics in past 90 days
* Willing to avoid taking probiotics during the study
* Has access to a safe place to perform aerobic exercise (e.g., willing to walk in neighborhood or has gym membership or owns relevant exercise equipment at home, etc.)
* Has access to good internet and WIFI and device capable of videoconferencing (the study has limited resources to loan tablets and hotspots)

Exclusion Criteria:

* Metastatic or recurrent cancer
* Another cancer diagnosis in the past 5 years (not including skin or cervical cancer in situ)
* Unstable angina
* New York Heart Association class II, III, or IV congestive heart failure
* Uncontrolled asthma
* Interstitial lung disease
* Current steroid use
* Told by a physician to only do exercise prescribed by a physician
* Dementia or organic brain syndrome
* Schizophrenia or active psychosis
* Connective tissue or rheumatologic disease
* Participating in >30 minutes of exercise on ≥3 days/week in the past six months
* Anticipate elective surgery, medication changes or antibiotics during the study
* Contraindication to ≥moderate intensity aerobic exercise
* Physical limitations that prevent engaging in ≥moderate intensity aerobic exercise
* Breastfeeding, pregnant or anticipate pregnancy during the study
* Plan to move residence during the study
* Plan to travel for more than 1 week during the study
* Anticipate trouble attending the weekly study videoconference calls
* History of bariatric surgery
* Body weight greater than 440 lbs
* Any social, psychological, or physical condition that interferes with the participant's ability to complete study activities or unduly increases study risk

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-01-22 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Feasibility - Recruitment | Baseline
  Number of participants excluded or not agreeing to participate will be measured
Feasibility - Adherence to study protocol activities | Throughout 10 week study period
  Feasibility measure (e.g. percent of assessments and intervention sessions completed
Feasibility - Attrition rates | Throughout 10 week study period
  Feasibility measure of the number of participants who dropout or are withdrawn
Feasibility - Adverse events | Throughout 10 week study period
  Feasibility measure of the number of adverse events recorded by staff during the study period
Feasibility - Participant satisfaction | At conclusion of 10 week study period
  Self-Administered survey given to the participant at the conclusion of the 10 week study period

SECONDARY OUTCOMES:
Accelerometer Measured Free-living physical activity (e.g., minutes of activity) | Baseline
  Motion sensor measures physical activity not observed during intervention activities
Accelerometer Measured Free-living physical activity (e.g., minutes of activity) | 5 weeks after baseline
  Motion sensor measures physical activity not observed during intervention activities
Accelerometer Measured Free-living physical activity (e.g., minutes of activity) | 10 weeks after baseline
  Motion sensor measures physical activity not observed during intervention activities
Body fat percentage analysis using a Tanita bioelectrical impedance analysis scale | Baseline
  Measurement of body fat percentage (0-100%) where a lower percentage is better.
Body fat percentage analysis using a Tanita bioelectrical impedance analysis scale | 5 weeks after baseline
  Measurement of body fat percentage (0-100%) where a lower percentage is better.
Body fat percentage analysis using a Tanita bioelectrical impedance analysis scale | 10 weeks after baseline
  Measurement of body fat percentage (0-100%) where a lower percentage is better.
Muscle mass analysis using a Tanita bioelectrical impedance analysis scale | Baseline
  Measurement of muscle mass (0 - max body weight in kilograms) where having more muscle mass can be considered positive.
Muscle mass analysis using a Tanita bioelectrical impedance analysis scale | 5 weeks after baseline
  Measurement of muscle mass (0 - max body weight in kilograms) where having more muscle mass can be considered positive.
Muscle mass analysis using a Tanita bioelectrical impedance analysis scale | 10 weeks after baseline
  Measurement of muscle mass (0 - max body weight in kilograms) where having more muscle mass can be considered positive.
Body Mass Index analysis using a Tanita bioelectrical impedance analysis scale | Baseline
  Measurement of height (m) and weight (kg) to assess body mass index, where a higher body mass index is worse.
Body Mass Index analysis using a Tanita bioelectrical impedance analysis scale | 5 weeks after baseline
  Measurement of height (m) and weight (kg) to assess body mass index, where a higher body mass index is worse.
Body Mass Index analysis using a Tanita bioelectrical impedance analysis scale | 10 weeks after baseline
  Measurement of height (m) and weight (kg) to assess body mass index, where a higher body mass index is worse.
Change in physical performance | Baseline
  Participants will complete a 2-minute step test measured by study staff through videoconference
Change in physical performance | 5 weeks after baseline
  Participants will complete a 2-minute step test measured by study staff through videoconference
Change in physical performance | 10 weeks after baseline
  Participants will complete a 2-minute step test measured by study staff through videoconference
Composition of gut microbiota as measured by fecal samples | Baseline
  Using standard diversity and taxa comparison metrics
Composition of gut microbiota as measured by fecal samples | 5 weeks after baseline
  Using standard diversity and taxa comparison metrics
Composition of gut microbiota as measured by fecal samples | 10 weeks after baseline
  Using standard diversity and taxa comparison metrics
Fatigue measured through fatigue specific questionnaire | Baseline
  Fatigue Symptom Inventory which contains 13 items (fatigue intensity = mean of 4 items, 1 to 10 scale; fatigue interference = mean of 7 items, 0 to 10 scale; 2 general fatigue items = 0 to 7 scale and 1 to 10 scale); higher score indicates greater fatigue
Fatigue measured through fatigue specific questionnaire | 5 weeks after baseline
  Fatigue Symptom Inventory which contains 13 items (fatigue intensity = mean of 4 items, 1 to 10 scale; fatigue interference = mean of 7 items, 0 to 10 scale; 2 general fatigue items = 0 to 7 scale and 1 to 10 scale); higher score indicates greater fatigue
Fatigue measured through fatigue specific questionnaire | 10 weeks after baseline
  Fatigue Symptom Inventory which contains 13 items (fatigue intensity = mean of 4 items, 1 to 10 scale; fatigue interference = mean of 7 items, 0 to 10 scale; 2 general fatigue items = 0 to 7 scale and 1 to 10 scale); higher score indicates greater fatigue
Depression and Anxiety measured through specific questionnaire | Baseline
  Hospital Anxiety and Depression Scale [HADS] which contains 14 items (depression = total of 7 items, 0 to 3 scale; anxiety = total of 7 items, 0 to 3 scale) higher scores indicate greater depression and/or anxiety
Depression and Anxiety measured through specific questionnaire | 5 weeks after baseline
  Hospital Anxiety and Depression Scale [HADS] which contains 14 items (depression = total of 7 items, 0 to 3 scale; anxiety = total of 7 items, 0 to 3 scale) higher scores indicate greater depression and/or anxiety
Depression and Anxiety measured through specific questionnaire | 10 weeks after baseline
  Hospital Anxiety and Depression Scale [HADS] which contains 14 items (depression = total of 7 items, 0 to 3 scale; anxiety = total of 7 items, 0 to 3 scale) higher scores indicate greater depression and/or anxiety
Sleep dysfunction measured through specific questionnaire | Baseline
  Pittsburgh Sleep Quality Index which contains 7 components (sleep dysfunction = total of 7 components, 0 to 3 scale) higher score indicates worse sleep quality
Sleep dysfunction measured through specific questionnaire | 5 weeks after baseline
  Pittsburgh Sleep Quality Index which contains 7 components (sleep dysfunction = total of 7 components, 0 to 3 scale) higher score indicates worse sleep quality
Sleep dysfunction measured through specific questionnaire | 10 weeks after baseline
  Pittsburgh Sleep Quality Index which contains 7 components (sleep dysfunction = total of 7 components, 0 to 3 scale) higher score indicates worse sleep quality
Pain measured through Patient Reported Outcomes Measurement Information System [PROMIS®] | Baseline
  PROMIS® is a set of person-centered measures that evaluates and monitors physical health in adults (T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population) a higher score (higher SD) indicates greater pain
Pain measured through Patient Reported Outcomes Measurement Information System [PROMIS®] | 5 weeks after baseline
  PROMIS® is a set of person-centered measures that evaluates and monitors physical health in adults (T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population) a higher score (higher SD) indicates greater pain
Pain measured through Patient Reported Outcomes Measurement Information System [PROMIS®] | 10 weeks after baseline
  PROMIS® is a set of person-centered measures that evaluates and monitors physical health in adults (T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population) a higher score (higher SD) indicates greater pain
Post-traumatic stress measured through specific questionnaire | Baseline
  Post-traumatic Stress Disorder Checklist (PCL) which contains 20 items (PTSD intensity = total of 20 items, 0 to 4 scale) higher score indicates greater PTSD
Post-traumatic stress measured through specific questionnaire | 5 weeks after baseline
  Post-traumatic Stress Disorder Checklist (PCL) which contains 20 items (PTSD intensity = total of 20 items, 0 to 4 scale) higher score indicates greater PTSD
Post-traumatic stress measured through specific questionnaire | 10 weeks after baseline
  Post-traumatic Stress Disorder Checklist (PCL) which contains 20 items (PTSD intensity = total of 20 items, 0 to 4 scale) higher score indicates greater PTSD

CONTACTS AND LOCATIONS:
Overall Officials: Laura Rogers, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to share participant data.